CLINICAL TRIAL: NCT02251730
Title: A Feasibility and Efficacy Study of Smoking Cessation Program in Head and Neck Cancer Patients Receiving Curative Radiation Therapy
Brief Title: Smoking Cessation in Head and Neck Cancer Patients Receiving Curative Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201406075RINC
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Head and Neck Neoplasms
Keywords: radiation therapy,Smoking pattern,head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refer for smoking cessation (Experimental): Refer for smoking cessation
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Smoking cessation — Refer for smoking cessation

SUMMARY:
To propose a feasibility study of introducing a smoking cessation program in head and neck cancer patients with planned radiotherapy. The study will feature the feasibility, safety, and efficacy of a prospective smoking cessation program during head and neck irradiation.

DETAILED DESCRIPTION:
Smoking during radiotherapy in head and neck cancers yields not only more radiotherapy acute and late complications but also poor clinical tumor response, poor local control, and poor overall survival. However, smoking cessation has not been included into the standard intervention in treating head and neck cancer patients in Taiwan. We propose a prospective study of introducing a smoking cessation program in head and neck cancer patients receiving radiotherapy. The study will feature the feasibility, safety, and efficacy of a prospective smoking cessation program during head and neck irradiation. The primary outcome is to test the feasibility of the smoking cessation intervention, and the secondary outcome is to test the efficacy of the intervention during radiotherapy on acute and late RT toxicities, tumor response, patterns of relapse, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Head and Neck Malignancy Stage I-IVB without distant metastasis
* Receiving five weeks or more of external beam radiotherapy
* Report smoking one or more cigarettes in the past 30 days or self-identify as a smoker
* KPS 70-100

Exclusion Criteria:

* Serious or unstable cardiac, renal, hypertensive, pulmonary, endocrine, or neurologic disorders, as assessed by the study-site physician
* A current diagnosis of major depressive episode or a history of psychosis, bipolar disorder, or seizure disorder
* Pregnancy or lactation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Successful smoking cessation at the end of radiotherapy, confirmed by CO breath test concentrations of 3 ppm or less. | 10 weeks
  The primary outcome was to test the feasibility of introducing a smoking cessation program in head and neck cancer patients undergoing radiotherapy. Smoking cessation status will be formally assessed by patient report and by carbon monoxide (CO) breath test. The status of tobacco abstinence will be confirmed by carbon monoxide breath test concentrations of 3 ppm or less.

SECONDARY OUTCOMES:
≥ Grade 3 acute and late adverse event | 2 years
  The secondary outcomes were to test the efficacy of smoking cessation during radiotherapy on acute and late radiation therapy toxicities, tumor response, patterns of relapse, and overall survival.
One- and two-year local-regional control rates | 2 years
  All patients will be evaluated by the treating physician once per week during treatment, and acute toxicities will be rated with CTCAE v4.0. All patients will be followed up every 2-3 months for the first 2 years, every 4 months for the third year, and every 6 months until recurrence or death. Late toxicities will be assessed with late morbidity scoring criteria of Radiation Therapy Oncology Group.
One- and two-year distant metastases-free survival rates | 2 years
  All patients will be evaluated by the treating physician once per week during treatment, and acute toxicities will be rated with CTCAE v4.0. All patients will be followed up every 2-3 months for the first 2 years, every 4 months for the third year, and every 6 months until recurrence or death. Late toxicities will be assessed with late morbidity scoring criteria of Radiation Therapy Oncology Group.
One- and two-year progression-free survival rates | 2 years
  All patients will be evaluated by the treating physician once per week during treatment, and acute toxicities will be rated with CTCAE v4.0. All patients will be followed up every 2-3 months for the first 2 years, every 4 months for the third year, and every 6 months until recurrence or death. Late toxicities will be assessed with late morbidity scoring criteria of Radiation Therapy Oncology Group.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ling-Yu Chen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan